CLINICAL TRIAL: NCT02052843
Title: Impact Evaluation of the Steps to Success Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRP699103
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steps to Success (Experimental): Steps to Success enhanced home visits-including instruction for both young mothers and fathers on contraception, comprehensive sex education, and the importance of adequate birth spacing, and accompanied by group sessions on adulthood preparation topics.
  Interventions: Behavioral: Steps to Success
- Traditional Healthy Families (Active Comparator): Traditional Healthy Families home visits which cover topics of parenting and child development
  Interventions: Behavioral: Traditional Healthy Families

INTERVENTIONS:
Behavioral: Steps to Success
  Arms: Steps to Success
Behavioral: Traditional Healthy Families
  Arms: Traditional Healthy Families

SUMMARY:
The evaluation will examine whether the Steps to Success enhanced home visits are more effective at delaying repeat pregnancies than are traditional Healthy Families home visits.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 14 to 21
* Pregnant, or have delivered a child in the last three months

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 595 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Subsequent pregnancy | 2-years post random assignment

SECONDARY OUTCOMES:
Subsequent pregnancy | 1-year post random assignment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, p, Study Director — Mathematica Policy Research
Locations (1):
- Healthy Families San Angelo, San Angelo, Texas, United States